CLINICAL TRIAL: NCT02182219
Title: A Phase I Open Label Dose Escalation Study of Continuous (Except on the Days of Chemotherapy Infusion) Oral Treatment With BIBF 1120 Together With Docetaxel and Prednisone in Patients With Hormone Refractory Prostate Cancer
Brief Title: Oral Treatment With BIBF 1120 Together With Docetaxel and Prednisone in Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.4
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — nintedanib

ARMS (1):
- BIBF 1120 (Experimental)
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120

SUMMARY:
The primary objective of this study was to determine the safety and Maximum tolerated dose (MTD) of BIBF 1120 combination therapy with docetaxel and prednisone in patients with hormone refractory prostate cancer. Secondary objectives were to characterise the pharmacokinetic profiles of BIBF 1120 and docetaxel and possible Pharmacokinetic (PK) interactions between BIBF 1120 and docetaxel and to obtain preliminary information on anti-tumour activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-proven metastatic prostate adenocarcinoma
2. Progression after hormonal therapy
3. Progressive disease as follows:

   * Increase of PSA > 5 ng/ml on two occasions despite castrate levels of testosterone before screening
   * AND/OR Progressive measurable disease (RECIST criteria)
   * AND/OR Progressive bone metastases (presence of new lesion(s) on a bone scan)
4. Life expectancy of at least three months
5. ECOG performance status ≤ 2
6. Patient written informed consent obtained prior to any trial procedures and that is consistent with ICH-GCP (International Conference on Harmonization - Good Clinical Practice) guidelines.

Exclusion Criteria:

1. Prior treatment for hormone refractory prostate cancer (HRPC) including chemotherapy, biologic response modifier therapy, or any investigational drug
2. Participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
3. Major injuries and surgeries within the past 4 weeks. Planned surgical procedures during the trial
4. Brain metastases
5. Radiotherapy superior to 30% of the medullar volume
6. Other malignancy diagnosed within the past 5 years (other than non-melanomatous skin cancer)
7. Gastrointestinal abnormalities that would interfere with intake or absorption of the study drug, such as a requirement for intravenous alimentation, prior surgical procedures affecting absorption, treatment for peptic ulcer disease within the last 6 months, active gastrointestinal bleeding unrelated to cancer (as evidenced by either hematemesis, or melena in the past 3 months and without endoscopic documented resolution), or malabsorption syndromes
8. Previous history of stroke, angor pectoris, ischemic cardiomyopathy, cerebral ischemia, arteritis in the past 6 months
9. Recent history of hemorrhagic or evolutive thrombotic event (including transient ischemic attacks) in the past 6 months
10. Patients who require full-dose anticoagulation or heparinization
11. Absolute neutrophil count (ANC) < 1,500/μl, platelet count < 100,000/μl, or hemoglobin < 8 mg/dL
12. Total bilirubin > upper limit of normal (ULN); alanine amino transferase (ALT) and/or aspartate amino transferase (AST) >1.5 X ULN
13. Serum creatinine > 1.5 mg/dL (> 132 μ mole/L, SI Unit equivalent)
14. Known or suspected active alcohol or drug abuse
15. Patients unable to comply with the protocol

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2007-04-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to day 126
Incidence and intensity of Adverse Events according to the Common Terminology Criteria for Adverse Events (version 3.0) associated with increasing doses of BIBF 1120 | up to 6 months

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) over the dosing interval τ following the first dose (AUC0-24) | up to 336 hours after drug administration
Incidence of prostate specific antigen (PSA) decline ≥ 50% from the baseline value | Baseline, up to day 126
Number of patients with an objective tumour response (Partial Response (PR), Complete Response (CR)) according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria | Baseline, day 15 of cycle 3 and at the end of cycle 6
Number of patients without signs of tumour progression (stable disease (SD)) according to RECIST criteria | Baseline, day 15 of cycle 3 and at the end of cycle 6
Change in Eastern Cooperative Oncology Group (ECOG) performance score | Baseline, up to day 156
AUC over the time interval from zero to the time of the last quantifiable drug concentration after the first dose (AUC0-tz) within the dosing interval τ | up to 336 hours after drug administration
AUC over the time interval from zero extrapolated to infinity (AUC0-∞) after the first dose | up to 336 hours after drug administration
Percentage of AUC0-∞ obtained by extrapolation (%AUCtz-∞) | up to 336 hours after drug administration
Maximum measured plasma concentration (Cmax) following the first dose | up to 336 hours after drug administration
Time from dosing to the maximum plasma concentration (tmax) following the first dose | up to 336 hours after drug administration
Terminal rate constant in plasma (λz ) | up to 336 hours after drug administration
Terminal half-life (t1/2) | up to 336 hours after drug administration
Mean residence time (MRTpo) after oral administration | up to 336 hours after drug administration
Apparent clearance (CL/F) | up to 336 hours after drug administration
Apparent volume of distribution during the terminal phase (Vz/F) | up to 336 hours after drug administration
Pre-dose plasma concentration immediately before administration | Days 2, 3, 8 and 15
Plasma concentration at 24 hours following the first (C24,1) dose | 24 hours after administration
Mean residence time (MRTiv) after i.v. administration | up to 336 hours after drug administration
Clearance (CL) after i.v. administration | up to 336 hours after drug administration
Apparent volume of distribution during the terminal phase (Vz) after i.v. administration | up to 336 hours after drug administration
Apparent volume of distribution at steady state (Vss) | up to 336 hours after drug administration

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com